CLINICAL TRIAL: NCT00005879
Title: A Phase II Clinical Trial of a Selective Estrogen Receptor Modulator (LY353381*HCl) in High Risk Women With Fine Needle Aspiration Cytologic Evidence of Hyperplasia
Brief Title: LY353381 in Preventing Breast Cancer in Women With Hyperplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Carol Fabian, MD, Director, Breast Cancer Prevention Unit, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KUMC-HSC-7264-97; CDR0000067918 (Registry Identifier: PDQ (Physician Data Query)); NCI-P00-0146 (Other: NCI); U01CA077165 (NIH)
Record Dates: First submitted 2000-06-02; First posted 2003-01-27 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — LY 353381

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Arzoxifene (Experimental): LY353381, 20 mg daily
  Interventions: Drug: arzoxifene

INTERVENTIONS:
Drug: arzoxifene — one tablet daily
  Other Names: LY353381
  Arms: Arzoxifene
Drug: Placebo — matched tablet dialy
  Arms: Placebo

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. The use of LY353381 may be an effective way to prevent the development of breast cancer in women who have hyperplasia.

PURPOSE: Randomized phase II trial to study the effectiveness of LY353381 in preventing breast cancer in women who have hyperplasia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine if LY353381 hydrochloride improves baseline cytology in women at high risk for breast cancer.
* Determine if this drug modulates other potential surrogate endpoint biomarkers or drug effect biomarkers.
* Determine if cytologic improvement is associated with initial presentation of the various stratification factors.
* Determine whether cytology is correlated with other potential surrogate endpoint biomarkers or drug effect biomarkers and whether change in cytology is correlated with change in the other biomarkers.
* Monitor the effects of this drug in terms of quality of life and women's health.

OUTLINE: This is a randomized, double-blind, multicenter study followed by an open-label study for both arms. Patients are stratified according to cytologic status (hyperplasia with atypia vs hyperplasia without atypia), mutation status (known carrier for BRCA1 or BRCA2 genes vs known not to be a carrier of mutant genes), menopausal status (premenopausal vs postmenopausal), estrogen-receptor status, and participating center. Patients are randomized to one of two treatment arms.

* Arm I: Patients receive oral LY353381 hydrochloride once daily for 6 months.
* Arm II: Patients receive oral placebo once daily for 6 months. Patients in both arms then receive oral LY353381 hydrochloride for an additional 6 months.

Quality of life is assessed at baseline and then at 6 and 12 months.

Patients are followed at 2 weeks and then annually for 5 years.

PROJECTED ACCRUAL: A total of 210-220 patients will be accrued for this study within 2.5-3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Current random fine needle breast aspiration (FNA) evidence of 1 of the following:

  * Hyperplasia with atypia
  * Hyperplasia without atypia but with a 10-year modified Gail risk of at least 4%
  * Hyperplasia without atypia but with a BRCAPRO risk of at least 25%
  * Hyperplasia without atypia but with a known mutation in BRCA1 or BRCA2
  * Hyperplasia without atypia but with a history of contralateral ductal carcinoma in situ or invasive breast cancer
* FNA must have been taken during days 1-14 of the menstrual cycle for premenopausal women
* Classified as ACR class I-III on mammogram with stepwedge within past 6 months If intact uterus and/or ovaries, must have color doppler transvaginal pelvic sonogram within past 6 months showing endometrial thickening no greater than 13 mm premenopausal or no greater than 8 mm postmenopausal

  * No ovarian cysts felt to be possibly or probably non-physiologic that have not resolved to gynecologist's satisfaction on repeat sonogram
* Must agree to have or have had genetic counseling and genetic testing performed for BRCA1 and BRCA2
* No active cancer (e.g., detectable disease)
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Any

Performance status:

* Not specified

Life expectancy:

* At least 12 months

Hematopoietic:

* Hemoglobin greater than 10 g/dL
* Granulocyte count greater than 1,000/mm^3
* No deficiencies in protein C, protein S, or antithrombin III
* No activated protein C resistance

Hepatic:

* Albumin greater than 3.0 g/dL
* Bilirubin less than 1.5 mg/dL
* AST less than 100 U/L
* Alkaline phosphatase less than 200 U/L

Renal:

* Creatinine less than 1.5 mg/dL

Cardiovascular:

* No history of deep venous thrombosis not related to trauma or pregnancy
* No severe coronary artery disease
* No history of prior stroke

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study
* No other active cancer
* No retinal vein thrombosis
* No concurrent severe poorly controlled migraine
* No factor V Leiden mutation carrier

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 12 months since prior immunotherapy

Chemotherapy:

* At least 3 months between completion of prior KUMC phase II difluoromethylornithine (DFMO) study and baseline aspiration
* At least 12 months since prior chemotherapy

Endocrine therapy:

* Must not have started or stopped hormone replacement therapy or oral contraceptives within 6 months of baseline aspiration
* Must continue all hormone replacement therapy and/or oral contraceptives that were being taken at time of baseline aspiration
* At least 12 months since prior tamoxifen, raloxifene, or other antihormonal therapy

Radiotherapy:

* At least 3 months since prior radiotherapy

Surgery:

* At least 6 months between prior oophorectomy and baseline aspiration

Other:

* At least 2 weeks since the start of other new medication that would be ingested for 1 or more months

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2000-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol J. Fabian, MD, Study Chair — University of Kansas
Locations (2):
- United States (2):
  - University of Kansas Medical Center, Kansas City, Kansas
  - U.S. Oncology Research, Inc., Dallas, Texas

IPD SHARING:
Plan to Share IPD: No
Global results will be published.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screen by random periareolar fine needle aspiration for presence of hyperplasia or hyperplasia with atypia.
Period: Overall Study
Arm/Group | Placebo | Arzoxifene
Started | 101 | 98
Completed | 93 | 88
Not Completed | 8 | 10
Not completed — Withdrawal by Subject | 8 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Arzoxifene | Total
Number analyzed (Participants) | 101 | 98 | 199
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.5 (7.1) | 46.7 (6.6) | 46.6 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 98 | 199
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 101 | 98 | 199
Height [Mean (Standard Deviation); unit: inches] | 64.8 (2.6) | 65.1 (2.4) | 65.0 (2.5)
Weight [Mean (Standard Deviation); unit: lb] | 156 (32) | 157 (40) | 156 (36)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.3 (5.5) | 26.0 (5.8) | 26.1 (5.6)
Menopause Status [Count of Participants; unit: Participants]
  Pre | 52 | 51 | 103
  Post | 49 | 47 | 96
Hormone Use [Count of Participants; unit: Participants]
  None | 66 | 69 | 135
  OC or HRT Use | 35 | 29 | 64
Age at Menarche [Mean (Standard Deviation); unit: years] | 12.78 (1.42) | 12.82 (1.45) | 12.79 (1.43)
Age at First Live Birth [Mean (Standard Deviation); unit: years] | 20.6 (10.4) | 20.2 (12.1) | 20.4 (11.2)
Prior Biopsy [Count of Participants; unit: Participants] | 17 | 17 | 34
Number relatives with Breast Cancer [Count of Participants; unit: Participants]
  0 Relatives | 23 | 27 | 50
  1 Relative | 53 | 52 | 105
  2 Relatives | 23 | 17 | 40
  3 Relatives | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Masood Score
Description: Change in the semi-quantitative score assigned by the designated cytopathologist.
  Range 6-24. Score represents increasing abnormality (i.e., worse appearance) Sum composite of 6 cytomorphological features, each scored as 1-4.
Time Frame: Baseline to 6 months
Population: Analysis is restricted to subjects that complete the initial 6-month portion of the trial, have a repeat random periareolar fine needle aspiration, and are thus evaluable for change in Masood score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Arzoxifene
Number analyzed (Participants) | 84 | 82
units on a scale | -1.1 (1.9) | -0.8 (2.1)

2. Primary Outcome: Number of Participants With Improvement From Baseline in Cytomorphologic Abnormality at 6 Months
Description: Change (improvement) in categorical descriptor of cytologic abnormality as assigned by the primary cytopathologist.
  Categories include: normal (non-proliferative), epithelial hyperplasia, epithelial hyperplasia with atypia.
Time Frame: Baseline to 6 months
Population: Analysis is restricted to subjects that complete the initial 6-month portion of the trial, have a repeat random periareolar fine needle aspiration, and are thus evaluable for change in cytomorphology category.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Arzoxifene
Number analyzed (Participants) | 84 | 82
Participants
  No Improvement | 53 | 52
  Improvement | 31 | 30

ADVERSE EVENTS:
Time Frame: Duration on study agent, nominally a maximum of 12 months.
Arm/Group | Placebo | Arzoxifene
Serious Adverse Events (participants affected / at risk) | 5/101 | 9/98
Other Adverse Events (participants affected / at risk) | 100/101 | 97/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=101) | Arzoxifene (N=98)
APPENDICITIS (Gastrointestinal disorders) | 2 (2) | 0 (0)
SLIPPED DISK (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OVARIAN CYST (Reproductive system and breast disorders) | 1 (1) | 1 (1)
ISCHEMIC COLITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
UTERINE DISORDER / MULTIPLE UTERINE FIBROIDS (Reproductive system and breast disorders) | 0 (0) | 1 (1)
ANGIOEDEMA (Vascular disorders) | 0 (0) | 1 (1)
DEEP VEIN THROMBOSIS RIGHT CALF (Vascular disorders) | 1 (1) | 0 (0)
RIGHT BIMALLEOLAR ANKLE FRACTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BILATERAL CATARACTS (Eye disorders) | 0 (0) | 1 (1)
ACUTE MYELOID LEUKEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
PRIMARY DCIS IN BREAST (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=101) | Arzoxifene (N=98)
Asthenia (General disorders) | 21 (33) | 35 (54) — Fatigue
Vasodilation (General disorders) | 33 (72) | 58 (74) — Hot flashes
Leg Cramps (Musculoskeletal and connective tissue disorders) | 16 (39) | 41 (55)
Sweating (Skin and subcutaneous tissue disorders) | 28 (59) | 63 (73)
Metrorrhagia (Reproductive system and breast disorders) | 20 (37) | 34 (37)
Urinary Frequency (Renal and urinary disorders) | 13 (22) | 23 (26)
Vaginitis (Reproductive system and breast disorders) | 19 (31) | 29 (37)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes